CLINICAL TRIAL: NCT01132820
Title: A Phase II Evaluation of Cediranib (Recentin; AZD2171, IND#72740, NSC# 732208) in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Cediranib Maleate in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02043; NCI-2011-02043 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0229J; CDR0000674008; GOG-0229J (Other: NRG Oncology); GOG-0229J (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Recurrent Uterine Corpus Carcinoma
MeSH Terms: interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive cediranib maleate PO daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cediranib Maleate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well cediranib maleate works in treating patients with endometrial cancer that has failed to respond to initial chemotherapy or has come back after surgery, radiation therapy, or other forms of treatment. Cediranib maleate may stop the growth of tumor cells by blocking proteins made by tumors that can stimulate growth of tumor cells as well as blood vessels in and around tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of cediranib (cediranib maleate) in patients with either persistent or recurrent endometrial carcinoma.

II. To determine the frequency and degree of toxicity of cediranib as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version (v.)4.0 in this cohort of patients.

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free survival and overall survival. II. To estimate the probability of response without restriction on the duration of response documentation since study enrollment.

TERTIARY OBJECTIVES:

I. To determine if the response to cediranib correlates with high-expression of its receptor targets (e.g., vascular endothelial growth factor receptor [VEGFR] [1, 2, 3] and platelet derived growth factor receptor [PDGFR]).

II. To determine if the response to cediranib correlates with high endogenous circulating plasma levels of VEGFA, low-levels of its endogenous inhibitor, soluble fms-related tyrosine kinase 3 (sFlt-1) (the truncated, circulating portion of VEGFR-1), or circulating tissue factor (TF) or circulating prostate apoptosis response-4 (Par-4), both potential markers of tumor progression.

III. To determine if a high-expression of VEGFA on pre-treatment tumor specimens correlates with response to cediranib.

IV. To determine if expression of phosphorylated mitogen activated protein kinase (ERK) 1 and 2, c-Jun, signal transducer and activator of transcription 3 (Stat3), protein kinase C (PKC), and phosphorylated ribosomal protein S6 (p70S6) kinase correlates with resistance or sensitivity to cediranib.

OUTLINE:

Patients receive cediranib maleate orally (PO) daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial carcinoma, which is refractory to curative therapy or established treatments; histologic confirmation of the original primary tumor is required

  * Patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, and transitional cell carcinoma
* All patients must have measurable disease; measurable disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1); measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST version 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG Phase III protocol or Rare Tumor protocol for the same patient population
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2; patients who have received two prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
  * Any other prior therapy directed at the malignant tumor must be discontinued at least three weeks prior to registration
* Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma; initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease according to the following definition: cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa

  * Note: Patients on this non-cytotoxic study are allowed to receive one additional cytotoxic chemotherapy regimen for management of recurrent or persistent disease, as defined above; however, due to the novel nature of biologic compounds, patients are encouraged to enroll on second-line non-cytotoxic studies prior to receiving additional cytotoxic therapy
* Patients must have NOT received any non-cytotoxic chemotherapy for management of recurrent or persistent disease; prior hormonal therapy is allowed
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN) or creatinine (Cr) clearance >= 60 ml/min
* Bilirubin less than or equal to 1.5 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) less than or equal to 2.5 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Neuropathy (sensory and motor) less than or equal to grade 1
* Urine protein creatinine (UPC) ratio must be < 1.0 gm

  * If UPC ratio >= 1, collection of 24-hour urine measurement of urine protein is recommended
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) =< 1.5 x ULN
* Patients must have an amylase and lipase =< ULN
* Patients must have a thyroid stimulating hormone (TSH) level and a free thyroxine (free T4) level within the institutional normal limits
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements as specified
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception

Exclusion Criteria:

* Patients who have had prior therapy with cediranib (AZD 2171) or other VEGF pathway-targeted therapy
* Patient with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with serious, non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to the first date of cediranib (AZD 2171) therapy
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy or any brain metastases
* Patients with clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension defined as systolic > 150 mmHg or diastolic > 100 mmHg despite optimized antihypertensive therapy
  * Myocardial infarction or unstable angina within 6 months of the first date of cediranib (AZD 2171) therapy
  * New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication; women who have received prior treatment with an anthracycline (including doxorubicin and/or liposomal doxorubicin) and have an ejection fraction < institutional lower limit of normal (LLN) will be excluded from the study
  * CTCAE grade 2 or greater peripheral vascular disease
  * History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of cediranib (AZD 2171) therapy
  * Mean corrected QT interval (QTc) > 500 msec or history of familial long QT syndrome
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Patients undergoing invasive procedures as defined below:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of cediranib (AZD 2171) therapy
  * Major surgical procedure anticipated during the course of the study
  * Minor surgical procedures, fine needle aspirates, or core biopsies within 7 days prior to the first date of cediranib (AZD2171) therapy
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bender, Principal Investigator — NRG Oncology
Locations (87):
- United States (87):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Saint Luke's Hospital-Warren Campus, Phillipsburg, New Jersey
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 6/7/2010 and suspended to accrual on 3/7/2011. The study reopened on 11/21/2011 and closed on 4/30/2012.
Groups:
- Cediranib: Cediranib (RECENTIN; AZD2171) will be administered PO 30 mg daily. Each 28 day period will be considered a cycle. Treatment will continue until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | Cediranib
Started | 53
Completed | 48
Not Completed | 5
Not completed — Ineligible: wrong cell type | 1
Not completed — Ineligible:Improper pre-protocol therapy | 1
Not completed — Ineligible:Inadequate pathology | 1
Not completed — Never treated | 1
Not completed — Inadequate data | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cediranib
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.5)
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0
  30-39 years | 0
  40-49 years | 3
  50-59 years | 10
  60-69 years | 20
  70-79 years | 12
  80-89 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Effects as Assessed by the National Cancer Institute CTCAE v. 4.0
Description: Adverse Events (Grade 3 or higher)
Time Frame: Up to 5 years
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Cediranib
Number analyzed (Participants) | 48
Participants
  Leukopenia | 0
  Thrombocytopenia | 0
  Neutropenia | 0
  Anemia | 3
  Other Investigations | 4
  Other Blood/Lymphatics | 1
  Cardiac | 1
  Ear and labyrinth | 0
  Endocrine | 0
  Eye | 0
  Nausea | 1
  Vomiting | 4
  Other Gastrointestinal | 16
  General and administration site | 13
  Hepatobiliary | 0
  Infections/infestations | 6
  Injury/poisoning | 0
  Metabolism/nutrition | 8
  Musculoskeletal/connective tissue | 3
  Neoplasms benign/malignant | 4
  Peripheral sensory neuropathy | 0
  Nervous system | 1
  Psychiatric | 1
  Renal/urinary | 3
  Reproductive/breast | 1
  Respiratory/thoracic/mediastinal | 4
  Skin/subcutaneous | 0
  Vascular disorders | 18

2. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by RECIST 1.1. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall response (OR) = CR + PR.
Time Frame: For diesease evaluated by physical examination, response was assessed prior to each cycle. CT scan or MRI if used to follow lesion for measurable disease every other cycle from enrollment until stopping study therapy. The average time on study is 3 mnths
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cediranib
Number analyzed (Participants) | 48
percentage of participants | 12.5 [6 to 23]

3. Primary Outcome: Progression-free Survival (PFS) = > 6 Months
Description: Number of participants who survived for at least 6 months. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v.1.0) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: For disease evaluated by physical examination, progression was assessed prior to each cycle. CT scan or MRI if used to follow lesion for measurable disease every other cycle. Evaluated from time of enrollment until progression or death, up to 5 years
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cediranib
Number analyzed (Participants) | 48
percentage of participants | 33.3 [22 to 46]

4. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years.
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cediranib
Number analyzed (Participants) | 48
months | 12.5 [6.6 to 16.7]

5. Secondary Outcome: Progression Free Survival
Description: Time until disease progression, death, or date of last contact.
Time Frame: Disease that can be assessed by physical exam should be evaluated every cycle. disease assessed by imaging should be evaluated every other cycle. Time frame to determine the date of progression is from the date of enrollment up to 5 years after enrollment
Population: All eligible and evaluable patients
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cediranib
Number analyzed (Participants) | 48
Months | 3.61 [2.46 to 5.22]

6. Secondary Outcome: Response Without Regard to the Time of Documented Response
Description: Complete and partial tumor response by RECIST 1.1
Time Frame: Tumor responses with time restriction starts at enrollment and goes to 6 months after enrollment or until pt. off study therapy,whichever occurs first. Without time restriction starts at enrollment,lasts until off study therapy, median duration = 2.63 mth
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cediranib
Number analyzed (Participants) | 48
percentage of participants | 12.5 [6 to 23]

7. Other Pre Specified Outcome: Expression of Phosphorylated ERK1 and 2, c-Jun, Stat3, PKC, and p70S6 Kinase
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Levels of Receptor Targets Such as VEGFR (1, 2, 3) and PDGFR
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Plasma Levels of Endogenous Circulating VEGFA, Levels of Its Endogenous Inhibitor, sFlt-1 (the Truncated, Circulating Portion of VEGFR-1), Circulating TF, and Circulating Par-4
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: VEGFA Expression on Pre-treatment Tumor Specimens
Description: High vs low expression.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment.
Arm/Group | Cediranib
Serious Adverse Events (participants affected / at risk) | 20/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib (N=48)
Anemia (Blood and lymphatic system disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Colonic Perforation (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Rectal Fistula (Gastrointestinal disorders) | 1
Peritoneal Necrosis (Gastrointestinal disorders) | 1
Ileal Obstruction (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Multi-Organ Failure (General disorders) | 1
Death Nos (General disorders) | 1
Lung Infection (Infections and infestations) | 1
Bladder Infection (Infections and infestations) | 2
Alanine Aminotransferase Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Confusion (Psychiatric disorders) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib (N=48)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 17
Sinus Bradycardia (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Chest Pain - Cardiac (Cardiac disorders) | 1
Middle Ear Inflammation (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Hypothyroidism (Endocrine disorders) | 14
Hyperthyroidism (Endocrine disorders) | 1
Endocrine Disorders - Other (Endocrine disorders) | 1
Eye Disorders - Other (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Blurred Vision (Eye disorders) | 3
Dry Eye (Eye disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Dry Mouth (Gastrointestinal disorders) | 8
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 33
Vomiting (Gastrointestinal disorders) | 15
Anal Hemorrhage (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 11
Rectal Hemorrhage (Gastrointestinal disorders) | 2
Oral Dysesthesia (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 14
Oral Hemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 5
Abdominal Distension (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 22
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2
Rectal Pain (Gastrointestinal disorders) | 1
Fecal Incontinence (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Esophageal Pain (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
General Disorders And Administration Site Conditio (General disorders) | 1
Pain (General disorders) | 10
Flu Like Symptoms (General disorders) | 1
Edema Limbs (General disorders) | 2
Edema Face (General disorders) | 1
Fatigue (General disorders) | 39
Fever (General disorders) | 3
Gait Disturbance (General disorders) | 1
Chills (General disorders) | 1
Gallbladder Pain (Hepatobiliary disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 2
Skin Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 10
Bruising (Injury, poisoning and procedural complications) | 3
Investigations - Other (Investigations) | 1
Weight Loss (Investigations) | 16
Platelet Count Decreased (Investigations) | 11
Lymphocyte Count Decreased (Investigations) | 1
Lipase Increased (Investigations) | 1
Inr Increased (Investigations) | 2
Hemoglobin Increased (Investigations) | 1
Creatinine Increased (Investigations) | 11
Cholesterol High (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 4
Blood Bilirubin Increased (Investigations) | 1
White Blood Cell Decreased (Investigations) | 11
Aspartate Aminotransferase Increased (Investigations) | 12
Alkaline Phosphatase Increased (Investigations) | 7
Alanine Aminotransferase Increased (Investigations) | 9
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypernatremia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 23
Acidosis (Metabolism and nutrition disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 15
Peripheral Motor Neuropathy (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Intracranial Hemorrhage (Nervous system disorders) | 1
Headache (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Depressed Level Of Consciousness (Nervous system disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 4
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 10
Hematuria (Renal and urinary disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Vaginal Pain (Reproductive system and breast disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Vaginal Dryness (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 2
Breast Pain (Reproductive system and breast disorders) | 1
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2
Skin Induration (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Thromboembolic Event (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 29
Hot Flashes (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less